CLINICAL TRIAL: NCT06120517
Title: The Relationship Between Low Back Pain and Pelvic Floor Muscle Strength, Urinary
Brief Title: The Relationship Between Lumbar Disc Herniation and Urinary Incontinence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Selver Soğan, Director, Sanko University
Other Study IDs: FztSelverSevalSogan
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: emg- biofeedback — EMG activity shows the electrical activity measured during striated muscle contraction. The electrical activity of the muscle is in microvolts (1 volt = 1,000,000μV). Biofeedback units usually produce audio or visual feedback depending on the amount of electrical activity. Recording the bio-electrical activity of the muscle is a practical indicator of its contractility.

SUMMARY:
The purpose of this research; To evaluate the relationship between low back pain and pelvic floor muscle strength, urinary incontinence, constipation and sexual dysfunction in female individuals with lumbar disc herniation. No study on this has been found in the literature.

Hypotheses of the study; Ho: ''There is no difference in terms of the relationship between low back pain and Pelvic Floor Muscle Strength, Urinary Incontinence, Constipation and Sexual Dysfunction in Female Individuals with Lumbar Disc Herniation.'' H1: ''There is a difference in terms of the relationship between low back pain and Pelvic Floor Muscle Strength, Urinary Incontinence, Constipation and Sexual Dysfunction in Female Individuals with Lumbar Disc Herniation.''

DETAILED DESCRIPTION:
Low back pain is a problem that is caused by overwork and impaired functional capacity. It has been observed that the source of low back pain is due to intervertebral disc pathologies at a rate of up to 39%. Lumbar disc herniation; Low back pain, manicure and numbness in fullness or cracks, muscle weakness, difficulty in moving, weakness, inability to hold places, pulling when sitting and deterioration in conditions, sudden stabbing pain in the waist area when coughing or sneezing, bursting of the herniated nucleus pulposus (nucleus pulposus). Lumbar disc herniation can be detected in non-symptomatic cases. Lumbar disc herniation, Protruded disc herniation (eccentric overflow is present; the annulus is intact), Extruded disc herniation (the nucleus has passed the ruptured annulus; however, there is still a connection with the nucleus formation at the disc borders.), Sequestered disc herniation (The residual piece has ruptured with the disc space and It is in the form of a free fragment.). One of the biggest causes of lower back pain is the weakness of the core muscles and their not being active at the right time. It is documented as a cylindrical shaped structure that provides the distance between the core, body, fillings and arms. The role of active, passive and normal structures in core stabilization can be sustained. Passive structures; bone, cartilage and connective tissues, and active structures consist of muscles. Core muscles in core stability; The respiratory muscles are the diaphragm, transversus abdominus muscle, multifidus muscle and pelvic floor muscles. These muscles create trunk and lumbo-pelvic stability and have a very important role in the muscular chain. In addition, it seems that the ability to remember sequences and the activation responses of these muscles are impaired or slowed down. It can cause dysfunction, especially in the transversus abdominus, multifudus and pelvic floor muscles.

The purpose of this research; To evaluate the relationship between low back pain and pelvic floor muscle strength, urinary incontinence, constipation and sexual dysfunction in female individuals with lumbar disc herniation. No study on this has been found in the literature.

Hypotheses of the study; Ho: ''There is no difference in terms of the relationship between low back pain and Pelvic Floor Muscle Strength, Urinary Incontinence, Constipation and Sexual Dysfunction in Female Individuals with Lumbar Disc Herniation.'' H1: ''There is a difference in terms of the relationship between low back pain and Pelvic Floor Muscle Strength, Urinary Incontinence, Constipation and Sexual Dysfunction in Female Individuals with Lumbar Disc Herniation.''

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Protruded and Extruded Lumbar Disc Herniation, Those who are between the ages of 18-55, BMI below 30 kg/m2

Exclusion Criteria:

* Trauma, Tumoral Causes - Cancer, Signs of neurological disease, Diabetus Mellitus, Hypertension etc. systemic disorder, Operated Disc Herniation, pregnancy, Those diagnosed with sequestered disc herniation

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Since urinary incontinence problem is more common in women, our research was planned to be conducted on female gender.
Study Population: Female individuals between the ages of 18-55 diagnosed with lumbar disc herniation will be included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire | 1 weeks
  Oswestry Low Back Pain Disability Questionnaire: This test is designed to obtain information about how much your back (or leg) complaint affects your daily life. It includes sections such as pain intensity, personal care (washing, dressing, etc.), lifting loads, walking, sitting, standing, sleep, sexual life (if applicable), social life, and travel. There are 6 sub-items in each section. The numbers next to the marked sub-items are added up. If there is more than 1 checked option in the same question, the highest value is taken. The maximum score is 50. The total score is calculated as = {[total score] /[(number of marked questions)x5]}x100. The validation of the Turkish version of the Oswestry Disability Index for patients with low back pain was made in our country in 2004 by Yakut, Düger, Öksüz, Yörükan, Üreten, Turan, Kardeşliği, Kiraz, Krd, Kayhan Yakut, Güler
Pelvic Floor Muscle Strength Measurement | 1 weeks
  It is the measurement of the electrical activity occurring during pelvic floor muscle contraction and relaxation using superficial electrodes and reflecting it on the screen with appropriate equipment. The active electrode can be applied to the perineal area at 2 and 7 o'clock, 3 and 9 o'clock, or 5 and 11 o'clock. The reference electrode is usually attached to the adductor muscle group or medial to the tuber ischii. If dual channels are to be used, electrodes are placed on the abdomen. When evaluating pelvic floor muscle activity, segments such as basal rest, tonic activity - slow twitch muscles, phasic activity - fast twitch muscles, endurance are evaluated. In sEmg analysis, values such as work average, rest average, release average, onset average, peak and minimum are recorded.
King Health Survey | 1 weeks
  It is a tool recommended by the European Clinical Practice Guidelines. It is a frequently used questionnaire to evaluate the quality of life of patients with incontinence, consisting of 32 items and two parts. It includes 7 subheadings consisting of multiple items in addition to two single-item questions such as general health status and impact on quality of life. These include: role limitations, physical limitations, social limitations, limitations in personal relationships, emotional problems, incontinence-related sleep and energy disorders, and severity measurements for incontinence. The second part is the 11-item Symptom Severity Scale, which evaluates the presence and severity of urinary symptoms. The score of the Symptom Severity Scale varies between 0 (best) and 30 (worst). For other survey areas, scores range from 0 (best) to 100 (worst). The Turkish reliability and validity of the survey was tested in 2015.
Constipation Severity Scale | 1 weeks
  There are 16 questions in total within the scope of the scale. It includes Large Intestinal Laziness, Fecal Obstruction and Pain subdimension. The score in the Large Intestinal Laziness dimension is between 0 and 29, the score in the Fecal Obstruction dimension is between 0 and 28, and the score in the Pain dimension is between 0 and 16. In this context, the lowest score that can be obtained is 0, while the highest score is 73. High scores from the scale indicate that the symptoms are at a serious level. The reliability and validity study of this scale was conducted in our country by Kaya and Turan in 2011.
Sexual Quality of Life Scale - Female | 1 weeks
  This scale is a six-point Likert type and consists of 18 items. Each item is expected to be answered considering your sexual life in the last four weeks. In evaluating the scale, an item is scored between 1 and 6 (1 = Completely agree, 2 = Largely agree, 3 = Partially agree, 4 = Partially disagree, 5 = Largely disagree, 6 = Strongly disagree). The score range that can be obtained from the scale varies between 18-108. In this point system, the total score received from the scale is converted to 100. To convert the total scale score to 100; It is stated that the formula (raw score taken from the scale -18)x100/90 should be used. For example, the scale score of an individual whose total raw score from the scale is 63 is converted to 100; (63- 18)x100/90=50. A high score from the scale indicates that the quality of sexual life is good. The validity and reliability study of the Turkish version of this scale was conducted in our country by Tuğut and Gölbaşı in 2010.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanko University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided